CLINICAL TRIAL: NCT02198690
Title: Randomized Trial of a Mammography Decision Aid for Women Aged 75 and Older
Brief Title: Trial of a Mammography Decision Aid for Women Aged 75 and Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mara Schonberg, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2014P000108; R01CA181357 (NIH)
Record Dates: First submitted 2014-07-16; First posted 2014-07-24 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer Screening
Keywords: Mammography, Older women, decision making

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mammography Decision Aid (Experimental): Development and pilot testing of the decision aid (DA) has been described previously. In brief, the DA is written at a 6th grade reading level and includes information on 1) breast cancer risk factors for women >75 years; 2) health/life expectancy; 3) likely outcomes if screened and not screened with mammography; 4) competing mortality risks; 5) breast cancer treatments; and 6) a values clarification exercise. The last page asks users their intentions of being screened on a 15-point validated scale and invites users to share this information with their clinician. PCPs whose patients are randomized to receive the DA will be sent a copy of the DA via email and a link to an optional training on using the DA (5 informational slides and a 3-minute video).
  Interventions: Other: Mammography decision aid
- Home safety pamphlet (Placebo Comparator): To reduce response bias and to compensate for the time and attention required by the intervention group to read the DA, patients in the control arm will be provided a two page pamphlet on home safety for older adults developed by the American Geriatrics Society (AGS) Foundation for Health in Aging. PCPs whose patients are randomized to the receive the home safety pamphlet, will be sent an email informing them that their patient will be coming in early to read health educational materials for older adults as part of a study. We otherwise do not plan any intervention for control group PCPs because we do not want to change their usual behavior. However, if PCPs in the control arm request a copy of the educational materials then we will email them a copy of the home safety pamphlet.
  Interventions: Other: Home safety pamphlet

INTERVENTIONS:
Other: Mammography decision aid
  Arms: Mammography Decision Aid
Other: Home safety pamphlet
  Arms: Home safety pamphlet

SUMMARY:
The aim of this study is to test whether an educational pamphlet on mammography designed for women aged 75 and older improves older women's decision-making around mammography screening. The investigators aim to show that the educational pamphlet improves older women's knowledge of the pros and cons or screening and leads to fewer women in poor health with short life expectancy being screened.

DETAILED DESCRIPTION:
Women aged 75 and older are the fastest growing segment of the US population and breast cancer incidence increases with age. However, none of the randomized trials of mammography screening included women >74 years and it is not known if mammography helps these women live longer. Increasingly, data suggest that women need around 10 year life expectancy to have a chance at a mortality benefit from being screened with mammography. Meanwhile, there are immediate harms to screening older women including: pain, anxiety, complications from tests after a false positive mammogram (e.g., breast biopsy), and overdiagnosis (finding tumors that otherwise would never have caused symptoms in one's lifetime). Overdiagnosis is particularly concerning since some older women experience significant complications from breast cancer treatment. Guidelines state that there is insufficient evidence to recommend mammography screening for women aged 75 years or older and encourage clinicians to discuss the uncertainty about the balance of benefits and harms with older women. Yet, few older women are informed of potential harms of mammography before being screened, likely because explaining such uncertainty can be challenging and time consuming.

To improve older women's understanding of the benefits and risks of mammography screening, investigators previously developed and pilot tested a pamphlet decision aid (DA) on mammography screening for women aged 75+ years. The pilot pretest/posttest trial of 45 women 75+ years found that the DA resulted in older women being more knowledgeable about the benefits and risks of mammography, clearer in their values, and fewer intended to be screened, especially those with <10 year life expectancy.

Investigators now propose a large cluster randomized controlled trial (RCT) of the DA, using primary care physician (PCP) as the unit of randomization, to definitively evaluate the DA's efficacy. The investigators aim to recruit 550 women 75-89 years from 100 PCPs who provide care at an academic primary care or geriatrics practice in Boston, three community practices in the Boston metro area, or at an academic internal medicine or family practice in North Carolina. Patient participants will either receive the DA (intervention arm) or an educational pamphlet on home safety for older adults (control arm). The investigators chose to use PCPs as the unit of randomization rather than individual patients because they anticipate that some patients will share the DA with their PCPs. Once PCPs are exposed to the DA for one patient they could change their approach to screening which could lead to contamination of the control group making it more difficult to show an effect of the DA.

Aims:

The investigators will examine and evaluate the impact of providing information on benefits and risks of mammography screening to women aged 75 and older on:

1. receipt of screening;
2. intentions of being screened;
3. knowledge of the pros and cons of being screened;
4. decisional conflict around screening;
5. preferred decision-making role around mammography (active vs. passive/shared with physician);
6. documented discussions by PCPs of the risks and benefits of mammography screening in participants' notes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking women
* Aged 75 to 89 years
* Scheduled for a routine visit or physical with their PCP in the next 4-12 weeks
* Women who have not had a mammogram in 6 months but have had one in 2 years.

Exclusion Criteria:

* Women who have it documented in their screening sheet that they have chosen to stop screening
* Women with a history of atypical ductal hyperplasia (ADH) or non-invasive or invasive breast cancer
* Women with dementia (on problem list/reported by PCP).
* Women without capacity for informed consent.
* Women that report <7th grade education (the reading level of study materials)
* Patients from PCPs that participated in the pilot or are study investigators.
* Women whose PCPs already had 25 patients participate in the study (the cap per PCP)

Ages: 75 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 541 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Receipt of mammography screening | 18 months
  The investigators chose receipt of screening as the primary outcome since they anticipate that implementation of the DA will require that the DA impacts mammography use, especially for women with short life expectancy. The investigators will follow women for 15 months to guarantee at least two years of data since their last mammogram (the upper bound of the recommended screening interval). Research staff will review primary care notes, radiology records, and screening sheets (mammograms performed outside the medical system are manually entered on screening sheets). Research staff will contact patients or an alternate if follow-up is not complete in the medical records.

SECONDARY OUTCOMES:
Screening intentions | follow-up interview within 1 week
  The investigators will use a validated 15-point scale to assess one's propensity to being screened. The investigators will categorize scores as 1-5 (yes), 6-10 (unsure), or 11-15 (no). The investigators will compare participants who respond with yes vs. those who are unsure or plan not to be screened.
Knowledge of the pros and cons of mammography screening | follow-up interview within 1 week
  11 questions (2 multiple choice and 9 true/false); 7 were adapted from other studies and 4 were developed based on the material in the decision aid. Correct answers will be summed.
Decisional Conflict Scale (DCS) | Follow-up interview within 1 week
  The DCS is a validated 16 item scale to measure uncertainty around a decision, whether one feels informed, clear about their personal values, and supported in their decision-making (Cronbach's alpha=0.78 to 0.92);scores range 0-100 and lower scores indicate less conflict.
Decision-making role | Follow-up interview within 1 week
  The Control Preferences Scale (CPS) is commonly used to assess patients' preferred involvement in decision-making. Research staff will categorize responses as active (patient made the final decision) versus passive too or shared with doctor.
Preparation for Decision-Making | Follow-up interview within 1 week
  The investigators will ask women in the intervention arm (DA group) this validated 10 item index to see if the DA prepared them to communicate with their clinician (Cronbach's alpha=0.92-0.96). For the control arm, the investigators will modify this index to ask participants how the pamphlet affects their thoughts around home safety.
Acceptability | Follow-up interview within 1 week
  The investigators will ask about length, clarity, and whether women found the materials anxiety invoking and/or whether they would recommend them to a friend. For the DA only, the investigators will ask if the material is balanced.
Anxiety | Follow-up interview within 1 week
  The investigators will examine whether the educational materials invoke anxiety using the short form of Spielberger State-Trait Anxiety Inventory.
Home safety | Follow-up interview within 1 week
  The investigators will ask both groups their intentions to perform several home safety measures (e.g., check hot water setting) to keep participants blinded to whether they were randomized to the intervention of interest.
Screening discussions | 18 months
  Research staff will review PCP notes up to 18 months after participation (in case patients choose to bring up screening at the next visit rather than the index visit) to see if PCPs documented a discussion on mammography. The investigators will categorize a woman as having received a balanced screening discussion if a note includes either: a) discussion of a limitation of screening or b) that mammography was discussed AND whether or not the patient chose to continue screening. To ensure the validity of coding of whether screening discussions occurred, at least 3 investigators will read the de-identified paragraphs of participants' records and code whether they think a balanced discussion occurred. Discrepancies will be adjudicated by consensus between investigators.
Home safety discussions | 18 months
  Research staff will review PCP notes up to 18 months after participation (in case patients choose to bring up screening at the next visit rather than the index visit) to see if PCPs documented a discussion on home safety (e.g., fall prevention tips). The investigators plan to assess both screening and home safety to keep chart abstractors blinded to the outcome of interest. To ensure the validity of coding of whether home safety discussions occurred, at least 3 investigators will read the de-identified paragraphs of participants' records and code whether they think a discussion occurred. Discrepancies will be adjudicated by consensus between investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Mara A Schonberg, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (4):
- United States (4):
  - Affiliated Physicians Group, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - University of North Carolina Medical Center, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schonberg MA, Kistler CE, Pinheiro A, Jacobson AR, Aliberti GM, Karamourtopoulos M, Hayes M, Neville BA, Lewis CL, Wee CC, Fagerlin A, Nekhlyudov L, Marcantonio ER, Hamel MB, Davis RB. Effect of a Mammography Screening Decision Aid for Women 75 Years and Older: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2020 Jun 1;180(6):831-842. doi: 10.1001/jamainternmed.2020.0440. PMID 32310288